CLINICAL TRIAL: NCT01717417
Title: Three Dimensional Movement Analysis of Maxillary Impacted Canine Using TADs: a Randomized Clinical Trial
Brief Title: Three Dimensional Movement Analysis of Maxillary Impacted Canine: a Randomized Clincial Trial
Status: Completed | Type: Observational
Sponsor: University of Genova (Other)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Marco Migliorati, Doctor, University of Genova
Other Study IDs: MVM1; GU-1 (Other: Genoa University)
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Complicated Impacted Tooth
Keywords: impacted canine; miniscrew; cone beam

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- group 1: Patient treated with Trans Palatal Arch as anchorage for canine traction
  Interventions: Device: TPA
- Group 2: Patient treated with miniscrew as anchorage for canine traction
  Interventions: Device: miniscrew

INTERVENTIONS:
Device: miniscrew
  Groups: Group 2
Device: TPA
  Groups: group 1

SUMMARY:
Maxillary canines are the second-most frequently impacted teeth in the dental arch after the third molars. The suspicion of a maxilary canine impaction raises with the absence of the permanent canine in the arch after the normal period of eruption, and has to be confirmed by a clinical evaluation of the patient and a radiographic assessment.

The approaches to the management of impacted canines are many, but the preferred approach typically involves surgical exposure and guided orthodontic eruption.

The initial mechanical eruption can be achieved in several ways, but an important distinction has to be done according to the anchorage method. The aim of this study is comparing Temporary Anchorage Devices (TADs), and cantilevers with a TMA sectional, using the quantification of canines and molars displacement as the main parameter.

A TAD is a mini screw temporarily fixed to bone for the purpose of enhancing orthodontic anchorage either by supporting the reactive unit (the anchoring tooth) or by obviating the need for it at large, and is subsequently removed after use.

The mini screw employed in this clinical trial will be an alloy type IV titanium screw with 1.5mm diameter and 8-10 mm long, and under local anesthesia will be placed in an area between the first premolar and first molar, on the buccal or labial side according to the canine position and teeth position.

For the evaluation of the canines and molar displacement, two CBCT will be required: the first one before the beginning of the traction (T0), the second one after three months (T1). Both the CBCT will be imported in the MIMICS image processing software (Materialize Group, Leuven, Belgium). Limiting the tissue density ranges and restricting the anatomical area of interest, a cropped colored mask will be obtained from each CBCT. Then the co-registration, through the identification of 5 at least landmark points, will allow the overlap of the two masks. At this point, calculating the 3D surface models, the tooth pre- and post-treatment positions will be evident and the measurement of the displacement possible.

ELIGIBILITY:
Inclusion Criteria:

* presence of one or two impacted maxillary canine requiring surgical exposure and orthodontic treatment

Exclusion Criteria:

* permanent teeth extraction-based treatment
* current or previous orthodontic treatment in the last 12 months
* current systemic disease
* current antibiotic or antinflammatory therapy that can may compromise the result

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients referred to the Orthodontic Department, Genoa University.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-14 (Actual)

PRIMARY OUTCOMES:
Canine movement | baseline and 3 months after starting treatment
  Superimposition of two consecutive TC cone beam using at least 5 landmarks point. Calculation of the 3D surface model and the measureament of the canine and first molar movement

SECONDARY OUTCOMES:
Side effect of traction | baseline and end of treatment
  Evaluation of Root cervical resorption of other teeth due to canine movement Bone density after three month of traction

CONTACTS AND LOCATIONS:
Overall Officials: Armando Silvestrini Biavati, MD, DDS, Study Director — Genoa University, Italy; Marco Migliorati, DDS, MSc, Principal Investigator — Genoa University, Italy
Locations (1):
- Orthodontics Department, Dental School, Genoa University. Italy, Genoa, Italy

REFERENCES:
- [Derived] Migliorati M, Cevidanes L, Sinfonico G, Drago S, Dalessandri D, Isola G, Biavati AS. Three dimensional movement analysis of maxillary impacted canine using TADs: a pilot study. Head Face Med. 2021 Jan 15;17(1):1. doi: 10.1186/s13005-020-00252-0. PMID 33451343